CLINICAL TRIAL: NCT00820274
Title: Evaluation of the Cryopreserved Amniotic Membranes in the Care of Resistant Vascular Ulcers
Acronym: MAUV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: clinical trial have encountered difficulties enrolling a sufficient number of patients
Sponsor: University Hospital, Limoges (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I07011
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2013-12

CONDITIONS: Resistant Vascular Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- amniotic membranes (Experimental)
  Interventions: Procedure: amniotic membranes

INTERVENTIONS:
Procedure: amniotic membranes — The amniotic membrane is taken with a sterile crowbar then applied side foetal face against the ulcer and displayed in a homogeneous way

SUMMARY:
To evaluate tolerance and efficiency of cryopreserved amniotic membranes in local treatment of resistant vascular ulcers.

To evaluate complete cicatrisation, efficiency on pain, prevention of infection, improvement of quality of life.

To evaluate rate of amputations and recurrence at one year after complete cicatrisation

DETAILED DESCRIPTION:
Treatment of patients suffering from vascular ulcers or amputation's wound from at least 6 months after or without possibility for surgical treatment. A cryopreserved amniotic membrane, obtained after caesarean from consenting women without any disease, is applied on the ulcer after serological checking and changed once a week.

Main criterias:

Tolerance will be evaluated on clinical criterias. Efficiency will be evaluated by measuring reduction of ulcer's area (reduction of at least 50 % at 6 months).

Secondary criterias:

Reduction of pain will be evaluated by analogic visual scale and evaluation of analgesic consumption.

Evaluation of infections, amputations, complete healing, improvement of quality of life by SF36 questionnaire and recurrence at one year for patients with complete healing.

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent
* Leg or foot arterial or mixed ulcer older than at least 3 months

Exclusion Criteria:

* No obtained informed consent
* Possibility for surgical treatment (revascularisation)
* Age less than 18
* Pregnancy
* Indication for major amputation (below /above the knee)
* Venous ulcer
* Ulcer with infection and / or necrosis
* Mycotic ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Measure of the diameter of the ulcer | Every week

CONTACTS AND LOCATIONS:
Overall Officials: Francis Pesteil, MD, Principal Investigator — CHU Limoges
Locations (3):
- France (3):
  - Service de Médecine Interne et Pathologie Vasculaire, Bordeaux
  - Service de Chirurgie Vasculaire et Viscérale, Bordeaux
  - Service de Chirurgie Thoracique, cardiovasculaire et angiologie, Limoges